CLINICAL TRIAL: NCT06470490
Title: Effect of Psycho-Educational Program and Relaxation Training on Resilience, Self- Esteem and Psychological Distress Among Women With Breast Cancer
Brief Title: Effect of Psycho-Educational Program and Relaxation Training on Resilience Among Women With Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abeer Abd Elwahed Almowafy (Other)
Responsible Party: Sponsor-Investigator, Abeer Abd Elwahed Almowafy, Clinical Professor, Al-Azhar University
Organization: Al-Azhar University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Assiut University
Record Dates: First submitted 2024-06-03; First posted 2024-06-24 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Women With Breast Cancer
Keywords: Self-esteem; Psychological Distress; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- a psychoeducational program and relaxation training (Experimental): a psychoeducational program and relaxation training
  Interventions: Behavioral: psychoeducational
- routine care without the psychoeducational program (No Intervention): routine care without the psychoeducational program

INTERVENTIONS:
Behavioral: psychoeducational — educational program
  Arms: a psychoeducational program and relaxation training

SUMMARY:
Aim: To evaluate the effect of psycho-educational program and relaxation training on resilience, self-esteem, and psychological distress among women with breast cancer.

Design: Randomized controlled trials used a pretest and posttest design to determine the effect of psychoeducational program and relaxation training on resilience, self-esteem, and psychological distress among women with breast cancer presenting to breast clinics in Assiut, Egypt. The women were randomly allocated to the intervention group and control group.

Method: Data collection took place at the outpatient clinic at the Assiut University in South Egypt Cancer Institute. The study involved a total of 100 participants diagnosed with breast cancer recruited using a purposive sampling method, who were categorized into two groups, each comprising 50 women. Group 1 received a psychoeducational program and relaxation training, while Group 2 received only routine care without the psychoeducational program. Inclusion criteria were age ranging from 20 to 60 years, consent to research participation, and nonmetastatic breast cancer diagnosis. The investigators excluded failing to engage regularly in the psychoeducational program, suffering from a significant illness other than breast cancer, having a history of persistent psychological illnesses, and using psychiatric medications.

DETAILED DESCRIPTION:
Breast cancer is the most frequent kind of cancer among women in developed as well as developing nations, and it is the leading malignancy among females in Egypt

ELIGIBILITY:
Inclusion Criteria:

* Age ranging from 20 to 60 years
* Consent to research participation
* Nonmetastatic breast cancer diagnosis

Exclusion Criteria:

* Failing to engage regularly in the psychoeducational programme
* Suffering from a significant illness other than breast cancer
* Having a history of persistent psychological illnesses
* Using psychiatric medications.

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 100 (Actual)
Dates: Start 2024-01-07 (Actual); Primary Completion 2024-03-14 (Actual); Study Completion 2024-05-02 (Actual)

PRIMARY OUTCOMES:
Measurement tool: questionnaire The psychoeducational intervention employed was effective in enhancing resilience and self-esteem while changing psychological distress among women diagnosed with breast cancer | 5 months
  The effect of psycho-educational program and relaxation training on resilience, self-esteem, and psychological distress among women with breast cancer

CONTACTS AND LOCATIONS:
Overall Officials: Saleh O Abdullah, prof, Study Director — Assiut
Locations (1):
- Faculty of Nursing, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No